CLINICAL TRIAL: NCT05725083
Title: Lower Thoracic Epidural Versus Erector Spinae Block for Postoperative Analgesia for Percutaneous Nephrolithotomy
Brief Title: Lower Thoracic Epidural vs Erector Spinae Block for PNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Keroles Heshmat Ghaly Seif, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Epidural vs ESPB in PCNL
Record Dates: First submitted 2023-01-25; First posted 2023-02-13 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Percutaneous Nephrolithotomy
Keywords: Lower thoracic epidural; Erector spinae block; Postoperative analgesia for PCNL

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower thoracic epiduarl (Experimental): before induction of anesthesia,first the investigators identify the correct targeted thoracic level. All epidural block will be performed under all aseptic precautions with a 17-gauge Tuohy needle and 19 G flex-tip catheters. Using the loss of resistance to saline technique, catheter will be inserted 4 cm into the epidural space and a suitable test dose will be administered to exclude intravascular or sub-arachnoid injection. Bupivacaine 0.25% of 7.5-12 ml volume will be given bolus through the epidural catheter then continuous infusion of bupivacaine 0.1% will be infused at a rate of 5 ml/h up to 15ml/h .for breakthrough pain patient controlled analgesia (PCA) using nalbuphine 1 mg bolus , 10 min lockout period . The catheter will be removed under complete aseptic precautions after 48 hrs.
  Interventions: Procedure: Lower thoracic epidural
- Erector spinae block (Experimental): before induction of anasthesia ,highfrequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T9 spinous process. A 21G 10 cm needle will be inserted using an in plane approach. The tip of the needle will be placed into the fascial plane on the deep aspect of the erector spinae muscle.confirmed by visible fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging.Then the catheter placement 5cm into the space under the erector spinae muscle and suitable test dose will be administered . Bupivacaine 0.25% of 7.5-12 ml volume will be given bolus through the catheter then continuous infusion of bupivacaine 0.1% will be infused at a rate of 5 ml/h up to 15 ml/h , for breakthrough pain patient controlled analgesia (PCA) using nalbuphine 1mg bolus,10 min lockout period.The catheter will be removed under complete aseptic precautions after 48 hrs.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Lower thoracic epidural — before induction of anesthesia,first the investigators identify the correct targeted thoracic level. All epidural block will be performed under all aseptic precautions with a 17-gauge Tuohy needle and 19 G flex-tip catheters. Using the loss of resistance to saline technique, catheter will be inserted 4 cm into the epidural space and a suitable test dose will be administered to exclude intravascular or sub-arachnoid injection. Bupivacaine 0.25% of 7.5-12 ml volume will be given bolus through the epidural catheter then continuous infusion of bupivacaine 0.1% will be infused at a rate of 5 ml/h up to 15ml/h .for breakthrough pain patient controlled analgesia (PCA) using nalbuphine 1 mg bolus , 10 min lockout period . The catheter will be removed under complete aseptic precautions after 48 hrs.
  Arms: Lower thoracic epiduarl
Procedure: Erector spinae plane block — before induction of anasthesia ,highfrequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T9 spinous process. A 21G 10 cm needle will be inserted using an in plane approach. The tip of the needle will be placed into the fascial plane on the deep aspect of the erector spinae muscle.confirmed by visible fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging.Then the catheter placement 5cm into the space under the erector spinae muscle and suitable test dose will be administered . Bupivacaine 0.25% of 7.5-12 ml volume will be given bolus through the catheter then continuous infusion of bupivacaine 0.1% will be infused at a rate of 5 ml/h up to 15 ml/h , for breakthrough pain patient controlled analgesia (PCA) using nalbuphine 1mg bolus,10 min lockout period.The catheter will be removed under complete aseptic precautions after 48 hrs.
  Arms: Erector spinae block

SUMMARY:
compare the efficacy of Lower Thoracic Epidural with Erector spinae plane block (ESPB) for post-operative analgesia after Percutaneous Nephrolithotomy with a hypothesis that both Lower Thoracic Epidural and Erector spinae plane block are effective in providing post-operative analgesia.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is the treatment of choice for patients with multiple or complex kidney or upper urinary tract stones, which necessitates the meticulous multi-modality analgesia due to mild to moderate pain originated from renal capsule dilation or nephrostomy-tube-related stress during the first 24 h after operation.

The main sources of the acute pain after PCNL are visceral pain originating from the kidneys and ureters, and somatic pain from the site incision. Renal pain is conducted through T10-L1 spinal nerves while ureter pain is conducted through T10-L2. Moreover, cutaneous innervation of the site of the incision is predominantly supplied by T10-T11 (T8-T12) because the incision site and tract for PCNL is usually used in the tenth to eleventh intercostal space, or in the subcostal area Blockade of both somatic and visceral nerves that innervate skin, muscle, kidneys, and ureters is required for the achievement of adequate analgesia after PCNL. Complete blockade of unilateral spinal nerves from T10 to L2 can provide sufficient analgesia during PCNL. This can be achieved by several regional techniques such as Lower Thoracic Epidural , Thoracic paravertebral block, Transversus abdominis block, Erector spinae block, and peri-tubal local anaesthetic infiltration .

PCNL surgery also has an increased risk for postoperative pulmonary complications because the procedure is performed near the diaphragm, especially, when approached through the upper pole of the kidney which increases the possibility of pleural and lung injuries. with poor control of the postoperative pain, this can result in decreased inspiratory and vital capacities and increase the incidence of lung atelectasis and postoperative hypoxemia. Multimodal analgesia techniques are utilized broadly to manage postoperative pain. The concept of multimodal analgesia implies not only providing analgesic drugs, but also performing nerve blocks with local anaesthetics.

Since Forrero et al. first described the Erector Spinae Plane Block (ESPB), the indications and clinical use of the block for different surgical interventions have been growing . Although, ESPB is an interfascial plane block, anatomical studies support the idea that some of its clinical benefit may derive from spread to the paravertebral and epidural space. Regional anesthesia may reduce the rate of chronic pain after surgery . Thoracic epidural blockade (TEB) using local anesthetic agents has been widely regarded as the gold standard for analgesia and reduction of associated complications following surgery.

Epidural analgesia was first accomplished by blockage with local anesthetics, and bupivacaine has been called the local anesthetic of choice for epidural infusion.. Epidural local anesthetics have been administered by continuous infusion in an attempt to minimize side effects , Nevertheless, hypotension as well as motor block , numbness , nausea and urinary retention have occurred.

Good analgesia from an epidural block can result in relieving postoperative pain , early extubation, better ventilatory mechanics and gas exchange and reduced rates of lung collapse, pneumonia and pain . However, the technique requires highly trained medical staff not only for insertion and removal of the epidural catheter but also for the management of the continuous infusion of pain medication. The risks associated with insertion of the epidural include accidental dural puncture, inadvertent high block, local anesthetic toxicity and total spinal anesthesia (inadvertent spinal injection of an epidural dose of local anesthetic), nerve injury, epidural hematoma and abscess are rare but serious complications.

Epidural is not a suitable technique for all patients and is contraindicated in patients with local infection, previous spinal surgery, disorders of blood clotting and in those taking anti-coagulant and anti-platelet therapy .

Thus, in the current study the investigators aim to compare the post-operative analgesic effect of Lower Thoracic Epidural with that of ESPB after Percutaneous Nephrolithotomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years with a body mass index (BMI) of 18-35 kg/m2
* patients with the American Society of Anesthesiologists (ASA) physical status I/II,
* Patients scheduled for elective Percutaneous Nephrolithotomy.

Exclusion Criteria:

* Contraindication to local anesthesia :

Allergy to local anaesthetics , Infection at the site of injection , Coagulopathy

* Chronic pain syndromes
* Prolonged opioid medication
* Patients who received any analgesic 24 h before surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption | 48 hours postoperatively
  Total opioid used

SECONDARY OUTCOMES:
First analgesic request | 48 hours postoperatively
  When the patient first time need analgesia
Pain scores | 48 hours postoperatively
  Numerical rating scale
Analgesic drug consumption other than Nalbuphine | 48 hours postoperatively
  Another drug needed and it's consumption
Ambulation Time | 48 hours postoperatively
  The time the patient first ambulated following the surgical procedure
Patient satisfaction with anathesia | 48 hours postoperativelyi
  If the patient feels pain using Visual Analogue Scale
Heart rate in beats per minute | Intraoperatively
  Heart rate be stable during operation
Mean arterial pressure in mmHg | Intraoperatively
  Be stable during operation
Incidence of postoperative nausea and vomiting | 48 hours
  If the patient feels vomiting and nausea and when
Block related complication | 48 hours postoperatively
  If there is any complications as local anesthetic toxicity , pneumothorax and vascular puncture during block procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mohamed Abd EL Latif, Professor, Study Chair — Assuit University Hospital; Amr Mohamed Ahmed Thabet, Lecturer, Study Director — Assuit University Hospital

REFERENCES:
- See also: Paravertebral block for surgical anesthesia of percutaneous nephrolithotomy — https://pubmed.ncbi.nlm.nih.gov/27428208/
- See also: abdominal wall blocks — https://pubmed.ncbi.nlm.nih.gov/28085788/
- See also: Thoracic paravertebral block for postoperative pain management in percutaneous nephrolithotomy patient — https://pubmed.ncbi.nlm.nih.gov/23257888/
- See also: Thoracic paravertebral block versus epidural anesthesia combined with moderate sedation for percutaneous nephrolithotomy — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5588437/
- See also: Percutaneous nephrolithotomy under a multimodal analgesia regime. — https://pubmed.ncbi.nlm.nih.gov/19397428/
- See also: Application of TAP block in laparoscopic urologic surgery: Current status and future directions. — https://pubmed.ncbi.nlm.nih.gov/30904960/
- See also: Pulmonary complications following percutaneous nephrolithotomy — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4024505/
- See also: Multimodal analgesia for controlling acute postoperative pain. — https://pubmed.ncbi.nlm.nih.gov/19606021/
- See also: The Erector Spinae Plane Block — https://pubmed.ncbi.nlm.nih.gov/27501016/
- See also: The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery — https://pubmed.ncbi.nlm.nih.gov/28272292/
- See also: Use of the ultrasound-guided erector spinae plane block in breast surgery — https://pubmed.ncbi.nlm.nih.gov/28492298/
- See also: Erector Spinae Plane Blocks Provide Analgesia for Breast and Axillary Surgery — https://pubmed.ncbi.nlm.nih.gov/29261601/
- See also: Continuous Erector Spinae Plane block for thoracic surgery in a pediatric patient — https://pubmed.ncbi.nlm.nih.gov/29226529/
- See also: Erector Spinae Plane Block Versus Retrolaminar Block — https://pubmed.ncbi.nlm.nih.gov/29794943/
- See also: A Cadaveric Study Investigating the Mechanism of Action of Erector Spinae Blockade. — https://pubmed.ncbi.nlm.nih.gov/29746445/
- See also: Local anaesthetics and regional anaesthesia for preventing chronic pain after surgery — https://pubmed.ncbi.nlm.nih.gov/23076930/
- See also: Epidural catheter analgesia for the management of postoperative pain. — https://pubmed.ncbi.nlm.nih.gov/3515598/
- See also: Analgesia in thoracic surgery — https://pubmed.ncbi.nlm.nih.gov/18953284/
- See also: Paravertebral block with ropivacaine 0.5% versus systemic analgesia for pain relief after thoracotomy — https://pubmed.ncbi.nlm.nih.gov/15919319/
- See also: A comparison of the analgesic efficacy and side-effects of paravertebral vs epidural blockade for thoracotomy — https://www.ncbi.nlm.nih.gov/books/NBK72557/
- See also: Efficacy of ultrasound-guided erector spinae plane block for analgesia after laparoscopic cholecystectomy — https://pubmed.ncbi.nlm.nih.gov/31822353/